CLINICAL TRIAL: NCT01827189
Title: Evaluation of the Comprehensive Primary Care Initiative
Brief Title: Staffing Patterns of Comprehensive Primary Care Practices
Acronym: cpc
Status: Completed | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: cpc32813
Record Dates: First submitted 2013-04-01; First posted 2013-04-09 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Medicare Expenditures and Hospital Use, All Conditions
Keywords: primary care, Medicare costs, hospitalizations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Comprehensive primary care practices: Comprehensive primary care practices are the intervention group.
  Interventions: Other: Comprehensive primary care
- Comparison practices: Comparison practices are the case-control group--the matched set of practices in a comparison area--whose patients' outcomes will be compared to those of intervention practices.

INTERVENTIONS:
Other: Comprehensive primary care — Practices participating in the comprehensive primary care initiative receive a monthly amount from Centers for Medicare and Medicaid Services for each attributed Medicare patient, plus technical support of a learning collaborative, and can share in any net savings generated.
  Groups: Comprehensive primary care practices

SUMMARY:
Examines staff size and composition of the 496 advanced primary care practices participating in CMS's comprehensive primary care initiative, in 7 regions (states or local areas) that were selected for the demonstration.

DETAILED DESCRIPTION:
Participating practices all have electronic health records, submitted applications to participate in this demonstration program designed to improve primary care practices, and were selected as the most advanced of the applicants in terms of use of health information technology and certification as a medical home or possessing features similar to those of a medical home. Participating practices will receive monthly payments from Centers for Medicare & Medicaid (CMS) for Medicare patients attributed to the practice, and from other payers in the market taht are participating in the initiative. The demonstration began in October 2012 and will continue for 4 years. This early paper focuses on describing these practices at the outset of the demonstration.

ELIGIBILITY:
Inclusion Criteria:

* All Medicare fee-for-service patients who receive the majority of their Evaluation and Management visits from one of the study practices.

Exclusion Criteria:

* none.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medicare patients enrolled in traditional Medicare who receive the majority of their Evaluation and Management visits from one of the study practices.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Medicare expenditures per year for patients attributed to the practice | Four years

SECONDARY OUTCOMES:
number of preventable hospitalizations | four years

OTHER OUTCOMES:
number of emergency room admissions | four years

CONTACTS AND LOCATIONS:
Overall Officials: Randall S Brown, PhD, Principal Investigator — Mathematica Policy Research

IPD SHARING:
Plan to Share IPD: No
not allowed; data belong to the federal government